CLINICAL TRIAL: NCT04584814
Title: Pilot Study of Using the Scare Respirator: Effect on Synchronicity, Respiratory Rate, Heart Rate, Oxygen Saturation, Neonatal-Infant Pain Scale (NIPS) and Sleep-wake Cycle on Amplitude Electroencephalography( aEEG)
Brief Title: Analyze Changes in Respiratory Rate When Using the Scare Respirator
Acronym: RESPSUS
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Pontificia Universidad Catolica de Chile (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Sequential | Masking: None | Purpose: Treatment
Other Study IDs: 180926007
Record Dates: First submitted 2020-08-21; First posted 2020-10-14 (Actual); Last update posted 2022-09-21 (Actual); Status verified 2022-03

CONDITIONS: Apnea of Newborn; Preterm Labor
Keywords: respiratory rate; scare ventilator; sleep wake cycle
MeSH Terms: conditions — Obstetric Labor, Premature

STUDY DESIGN:
Intervention Model Description: 10 preterms are going to be put on random measures in 2 hours blocks of, no intervention 2 hours of scare ventilator settled at 20 cycles per minute, and 2 hours of scare ventilator at 40cycles per minute
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: Yes | US Export: Yes

ARMS (1):
- Babies born Preterm (Experimental): Preterm babies, healthy at the time of the study, free of neonatal diseases and/or sequelae or malformations or genetic diseases. They were random assigned to two-hours blocks of basal, and dorsal stimulation protocol at 20 or 40 times per minute, each.
  Interventions: Device: No intervention; Device: scare ventilator at 20; Device: scare ventilator at 40

INTERVENTIONS:
Device: No intervention — Basal analysis
Device: scare ventilator at 20 — To set scare ventilator by 20 cycles per minute
Device: scare ventilator at 40 — To set scare ventilator by 40 cycles per minute

SUMMARY:
Pilot study of 10 preterm, who are going to be randomly placed to 3 phases : 2 hour of basal observation of respiratory rate, heart rate, saturation, NIPS and aEEG recording, 2 hours with a 20cycles/minute with "scare ventilator", and 2 hours of 40 cycles/minute with "scare ventilator"

DETAILED DESCRIPTION:
With this pilot study the investigator's want to see if the "scare respirator" can modify the vital signs of the newborn (NB) and if there is a relationship according to the frequency per minute given by the scare respirator and the patient's respiratory rate.

The "scare respirator" has been used many times to prevent central apnea in the newborn. This involves using a mechanical ventilator, but instead of connecting it to the patient's trachea to inflate his lungs, the air flow is connected to a surgical glove that inflates and deflates, with the optimal respiratory rate that the patient should have. This will be placed on the back to stimulate it tactically giving the necessary impulse of inspiration so that the patient alone can acquire the movement.

The importance of the development of this study is that it has been seen that the "scare respirator" could avoid central apneas, but no studies have been done on the change in respiratory rate that occurs with the device or if it bothers the NB or alters its wakefulness sleep pattern.

It is intended to evaluate 10 premature infants, during 3 observation periods. Heart rate (HR), Respiratory rate (RR) and saturation, pain scale and aEEG sleep wake pattern will be evaluated; first a rest period between feeds as baseline, then with a scare respirator at 20 cycles per minute and finally at 40 cycles per minute. The differences of qualitative and quantitative variables will be assessed with ad-hoc statistical tests.

ELIGIBILITY:
Inclusion Criteria:

* hospitalized healthy preterm babies,
* weighing more than 1500g at the time of the study

Exclusion Criteria:

* babies receiving any respiratory support
* carrier of any mayor malformation or genetic condition

Ages: 1 Day to 1 Month | Sex: All | Healthy Volunteers: Yes
Age Groups: Child
Enrollment: 10 (Actual)
Dates: Start 2020-03-01 (Actual); Primary Completion 2021-10-31 (Actual); Study Completion 2022-03-01 (Actual)

PRIMARY OUTCOMES:
Change of respiratory Synchronicity with the scare ventilator between 20 and 40 cycles per minute (cpm) | ten minutes after each intervention starts and every ten minutes for 2 hours straight
  % of time were respiratory rate is synchronised with the scare ventilator input, two tales of statistical differences, at 20 and 40 cycles per minute (cpm)

SECONDARY OUTCOMES:
Change from baseline newborn HR using the scare ventilator at 20 cpm | pre-intervention, ten minutes after intervention starts and every ten minutes for 2 hours straight
  differences in HR mean with two tales of statistical analysis ,between the two study periods
Change from baseline newborn HR using the scare ventilator at 40 cpm | pre-intervention, ten minutes after intervention starts and every ten minutes for 2 hours straight
  differences in HR mean with two tales of statistical analysis ,between the two study periods
Change from baseline on Sleep-wake cycles (SWC) using the scare ventilator at 20 cpm | pre-intervention, ten minutes after intervention starts and every ten minutes for 2 hours straight
  % of time of aEEG SWC presence, two tales of statistical differences, between the 2 study periods
Change from baseline on Sleep-wake cycles (SWC) using the scare ventilator at 40 cpm | pre-intervention, ten minutes after intervention starts and every ten minutes for 2 hours straight
  % of time of aEEG SWC presence, two tales of statistical differences, between the 2 study periods
Change from baseline on Discomfort scale using the scare ventilator at 20 cpm | pre-intervention, ten minutes after intervention starts every ten minutes for 2 hours straight
  Differences with the NIPS average, two tales of statistical differences, between the two study periods (scale 0-12; 0-2 no pain, 3-4 moderate pain, 5 or more severe pain)
Change from baseline on Discomfort scale using the scare ventilator at 40 cpm | pre-intervention, ten minutes after intervention starts every ten minutes for 2 hours straight
  Differences with the NIPS average, two tales of statistical differences, between the two study periods (scale 0-12; 0-2 no pain, 3-4 moderate pain, 5 or more severe pain)
Change from baseline on RR using the scare ventilator at 20 cpm | pre-intervention, ten minutes after intervention starts every ten minutes for 2 hours straight
  differences in RR mean with two tales of statistical differences between the two periods
Change from baseline on RR using the scare ventilator at 40 cpm | pre-intervention, ten minutes after intervention starts every ten minutes for 2 hours straight
  differences in RR mean with two tales of statistical differences between the two periods
Change from baseline on oxygen saturation using the scare ventilator at 20 cpm | pre-intervention, ten minutes after intervention starts every ten minutes for 2 hours straight
  differences in mean oxygen saturation expressed as a % , with two tales of statistical differences between the two periods
Change from baseline on oxygen saturation using the scare ventilator at 40 cpm | pre-intervention, ten minutes after intervention starts every ten minutes for 2 hours straight
  differences in mean oxygen saturation expressed as a % , with two tales of statistical differences between the two periods

CONTACTS AND LOCATIONS:
Overall Officials: Paulina Toso, MD, Principal Investigator — Pontificia Universidad Catolica de Chile
Locations (1):
- Puc, Nicu, Santiago, Santiago Metropolitan, Chile